CLINICAL TRIAL: NCT06353165
Title: A Clinical Study to Investigate Stannous Fluoride Toothpaste on Antibacterial Effects in the Different Regions of the Mouth as Compared to Colgate Cavity Protection Toothpaste
Brief Title: Anti-bacterial Clinical Study on Teeth, Tongue, Cheek, Gum, and Saliva
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CRO-2022-12-BAC-SNF-THA-YPZ
Record Dates: First submitted 2024-03-03; First posted 2024-04-08 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Plaque, Dental
Keywords: bacteria; plaque; saliva
MeSH Terms: conditions — Dental Plaque; Plaque, Amyloid

STUDY DESIGN:
Intervention Model Description: blinded
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (Active Comparator): toothpaste brushing 2/day for 2 minutes
  Interventions: Drug: Colgate Dental Cream
- Group II (Experimental): toothpaste brushing 2/day for 2 minutes
  Interventions: Drug: Stannous fluoride toothpaste

INTERVENTIONS:
Drug: Stannous fluoride toothpaste — product containing 0.45% stannous fluoride
  Other Names: experimental
  Arms: Group II
Drug: Colgate Dental Cream — product containing 0.76% sodium monofluorophosphate
  Other Names: control
  Arms: Group I

SUMMARY:
This 4-week clinical study was designed to examine the antibacterial efficacy of brushing with a 0.454% stannous fluoride toothpaste with potassium nitrate and pyrophosphate compared to a toothpaste containing 0.76% MFP (marketed as Colgate Cavity Protection Toothpaste) in different regions of the mouth (dental plaque, tongue, cheek, gum surface and in saliva) 12 hours post-brushing (overnight) after 2 and 4 weeks of product use.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ages 18-70, inclusive.
* Subject is available during study duration and has no allergies to oral hygiene formulations.
* A minimum of 20 natural teeth with facial and lingual scorable surfaces.
* A willingness to read, understand, and sign the Informed Consent Form after the nature of the study has been fully explained to them. Subject should demonstrate a willingness to comply with all study procedures and clinical examination schedules.
* Subjects with a baseline whole mouth scores of dental plaque of 1.5 or more [Turesky Modification of Quigley-Hein] and gingivitis index of 1.0 or more [Loe-Silness].

Exclusion Criteria:

* Participation in any other clinical study or test panel including clinical studies with oral hygiene formulations within the one month prior to entry into the study.
* History of dental prophylaxis or treatments in the past month or during study duration.
* History of medical treatments including antibiotic, anti-inflammatory or anticoagulant therapy during the month preceding study enrollment.
* Subjects scheduled for medical procedures for the duration of the study.
* Difficulty complying with study procedures and examinations such as excessive gagging during oral assessment etc.
* History of significant adverse effects following use of oral hygiene products such as toothpastes and mouthrinses. Allergy to personal care/consumer products or their ingredients.
* History of diabetes or hepatic or renal disease, or medical or inflammatory conditions or transmittable diseases, e.g. heart disease or AIDS.
* History of rheumatic fever, heart murmur, mitral valve prolapse or other conditions requiring prophylactic antibiotic coverage prior to invasive dental procedures.
* Oral soft tissue pathology.
* History of active or severe periodontal disease and loose teeth.
* Gross dental caries, severe generalized cervical abrasion and/or enamel abrasion, large fractured or temporary restorations (based on visual examinations).
* Fixed or removable orthodontic appliance or removable partial dentures.
* Self-reported pregnancy or lactation.
* Subjects known to be an alcoholic, or a recovering alcoholic.
* History or current use of recreational drugs or other habit promoting products.
* Use of phenolic flavored products, such as mint flavored candies and chewing gum, during the study period.
* Ability to refrain from oral hygiene for twelve (12) hours prior to scheduled visit.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-03-08 (Actual); Primary Completion 2023-04-12 (Actual); Study Completion 2023-04-12 (Actual)

PRIMARY OUTCOMES:
Whole mouth scores of dental plaque | baseline, 2 week & 4 week
  Measuring the dental plaque using the Turesky Modification of Quigley-Hein.Subjects presenting with whole mouth scores for dental plaque of 1.5 or more [Turesky Modification of plaque will be enrolled.
  Quigley-Hein.
Measurement of total bacterial counts on tongue | baseline, 2 week & 4 week
  Scrapings from the surface of the tongue. All collected samples will be placed in sterile vials, labeled with subject information and transferred to the laboratory for analysis
Measurement of total bacterial counts on cheek | baseline, 2 week & 4 week
  Scrapings from the surface of the cheek mucosa. All collected samples will be placed in sterile vials, labeled with subject information and transferred to the laboratory for analysis
Measurement of gingivitis | baseline, 2 week & 4 week
  Using the Loe-Silness index.Subjects presening will 1.0 or more for gingivitis [Loe-Silness] will be enrolled.
Measurement of total bacterial counts in saliva | baseline, 2 week & 4 week
  Collected samples in saliva will be placed in sterile vials, labeled with subject information and transferred to the laboratory for analysis

CONTACTS AND LOCATIONS:
Locations (1):
- M U International Oral Science Research, Ltd., Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No